CLINICAL TRIAL: NCT02529631
Title: Randomized, Double-blind, Clinical Investigation to Compare Orlistat 60 mg and a Customized Polyglucosamine, Two Treatment Methods for the Management of Overweight and Obesity
Brief Title: RCT to Compare Orlistat and Polyglucosamine for the Management of Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 003/07
Record Dates: First submitted 2015-07-24; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Overweight; Obesity
Keywords: Polyglucosamine; L 112; overweight,; obesity; orlistat; weight reduction
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: orlistat 60mg capsules (Active Comparator): A tailored blister-strip for one day contains
  * three capsules with orlistat 60mg Administration: 3 times daily 1 capsule with each meal containing fat concomitant with
  * six placebo tablets Administration: 3 times daily 2 tablets with each main meal
  Interventions: Drug: orlistat 60 mg
- Medical device: polyglucosamine (Active Comparator): A tailored blister-strip for one day contains
  * three placebo capsules Administration: 3 times daily 1 capsule with each meal containing fat concomitant with
  * six tablets Administration: 3 times daily 2 tablets (whereas the 2 tablets in the mold "breakfast" are placebo tablets and the remaining 4 tablets for lunch and dinner contains poliglucosamine
  Interventions: Device: polyglucosamine

INTERVENTIONS:
Drug: orlistat 60 mg — In order to have comparable calorie intakes, all participants followed the recommendations of the German clinical practice guidelines on the management and prevention of obesity.
  Due to the different appearance of tablets and capsules, a double dummy design was chosen, a blister strip for each day and each participant had to take the same amount of capsules and tablets per day. The content of the blister strips: three orlistat 60 g capsules plus six placebo tablets.
  Arms: Drug: orlistat 60mg capsules
Device: polyglucosamine — In order to have comparable calorie intakes, all participants followed the recommendations of the German clinical practice guidelines on the management and prevention of obesity.
  Due to the different appearance of tablets and capsules, a double dummy design was chosen, a blister strip for each day and each participant had to take the same amount of capsules and tablets per day. The content of the blister strips: three blue placebo capsules plus two placebo tablets (morning) and four polyglucosamine tablets (noon and evening).
  Arms: Medical device: polyglucosamine

SUMMARY:
This trial compares two treatment methods:

1. Orlistat 60 mg to be taken three times daily one capsule; indicated for weight loss in overweight adults. Important is also that it is taken along with a reduced-calorie and low-fat diet.
2. Polyglucosamine tablets to be taken two times daily two tablets, taken with the two main meals with the highest fat content, indicated for weight maintenance and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 28 kg/m² and < 45 kg/m²
* Waist circumference > 80 cm (women) > 94 cm (men)

Exclusion Criteria:

* Energy intake lower than the standard value according to Miffin St-Jeor equation
* Pregnancy or breast-feeding
* Addiction to alcohol
* Inability to fulfil the requirement of the trial protocol
* Cancer ,malignant tumour
* Hypersensitivity reactions to crustaceans or ingredient of the study medication
* Chronic diseases not under control with adequate therapy
* Diabetes

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of participants in both groups with a weight reduction of >= 5 per cent compared to the initial weight. | 12 weeks

SECONDARY OUTCOMES:
BMI reduction | 12 weeks
  Achieved change of the BMI (cm/m²) of all participants in each group compared to the initial average BMI
Waist circumference reduction | 12 weeks
  Achieved change of the waist circumference of all participants in each group compared to the initial average WC

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Stoll, MD, Principal Investigator — Diabetological centre, Dreieich, Germany; Umberto Cornelli, MD, Principal Investigator — CorCon, Mailand, Italy
Locations (2):
- Diabetological Center, Dreieich, Hesse, Germany
- MAP Center, Rende, Cosenza, Italy

REFERENCES:
- [Derived] Stoll M, Bitterlich N, Cornelli U. Randomised, double-blind, clinical investigation to compare orlistat 60 milligram and a customized polyglucosamine, two treatment methods for the management of overweight and obesity. BMC Obes. 2017 Jan 11;4:4. doi: 10.1186/s40608-016-0130-4. eCollection 2017. PMID 28097013